CLINICAL TRIAL: NCT00970047
Title: Development of a Noninvasive Fetal Sex Determination Test Between 6 and 16 Weeks of Gestation
Brief Title: Development of a Fetal Sex Assay From Maternal Whole Blood
Status: Completed | Type: Observational
Sponsor: Sequenom, Inc. (Industry)
Responsible Party: Allan Bombard / Chief Medical Officer, Sequenom, Inc.
Other Study IDs: SQNM-FS-101
Record Dates: First submitted 2009-08-31; First posted 2009-09-02 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2009-10

CONDITIONS: Fetal Sex Determination
Keywords: pregnant; fetal sex determination; gender determination; noninvasive test; fetal DNA

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and PBMCs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant females: Women who are pregnant and between 6 and 16 weeks of gestation and who are 18 to 64 years of age.

SUMMARY:
Whole blood from pregnant women will be collected to develop a noninvasive fetal sex test.

DETAILED DESCRIPTION:
This is an observational study whereby samples will be tested to determine the presence or absence of fetal Y chromosome genes to test for the fetal sex of the baby. The blood draw will occur between 6 to 16 weeks of gestation. The fetal gender will be requested at or soon after delivery if fetal sex was not previously obtained by CVS or amniocentesis genetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-64 years of age
* Subject is female
* Subject is pregnant and between 6 and 16 weeks of gestation
* Subject provides a signed and dated informed consent
* If subject undergoes a routine ultrasound between weeks 16 and 28, she agrees to provide the fetal sex results
* If subject undergoes an invasive procedure, she agrees to provide the fetal sex results

Exclusion Criteria:

* None

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women between 6 and 16 weeks of gestation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2008-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Bombard, MD, MBA, Study Director — Sequenom, Inc.
Locations (3):
- United States (3):
  - NCOG Medical Group, San Diego, California
  - IGO, San Diego, California
  - Scripps Clinic Medial Group, San Diego, California